CLINICAL TRIAL: NCT03169829
Title: Safety and Efficacy of Plant-based Diets in Hemodialysis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-00455
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Renal Disease
Keywords: Hemodialysis; Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodialysis Patients (Experimental): Phosphorus and potassium homeostasis will be assessed based on the concentrations of phosphorus and potassium in blood samples collected in fasting, post-prandial, mid-afternoon, pre-dialysis states, as well as the concentrations of phosphorus-regulatory factors, calcitriol, parathyroid hormone and fibroblast growth factor-23. The participants will be transitioned gradually to a plant-rich diet
  Interventions: Dietary Supplement: Standard Diet; Dietary Supplement: Low-k; Dietary Supplement: Standard

INTERVENTIONS:
Dietary Supplement: Standard Diet — Adapted from National Kidney Foundation guidelines for HD1
  * Animal only Protein
  * Refined only Grains
  * Limit Dairy
  * Low-k only
Dietary Supplement: Low-k — •¼ Animal, ¾ Plant Proteins
  •½ Refined, ½ Whole Grain
  * Limit Dairy, provide Soymilk Dairy
  * Low-k only Fruit and Vegetables
Dietary Supplement: Standard — •¼ Animal, ¾ Plant Proteins
  * Refined, ½ Whole Grain
    •Limit Dairy, provide Soymilk Dairy
  * Low-k, Fruit and Vegetables
  * High-k Fruit and Vegetables

SUMMARY:
The purpose of this proof-of-concept controlled-feeding study is to evaluate the impact of plant-rich diets, with and without high-potassium fruits and vegetables, on phosphorus and potassium homeostasis in hemodialysis (HD) patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving thrice-weekly outpatient HD treatments for end-stage renal disease
* 3-month mean serum potassium and phosphorus concentrations of >4.5 mEq/L and >4.0 mg/dL, respectively
* No prior episodes of moderate-severe hyperkalemia (potassium ≥6.5 mEq/L) in the past 6 months
* Deemed appropriate for the intervention by the patient's nephrologist, considering the patient's prognosis, cognition and pending treatments (e.g., kidney transplant)

Exclusion Criteria:

* Change in medications that alter potassium homeostasis (e.g., RAAS inhibitors, diuretics, beta-blockers) in the last month
* Diagnosed with bowel diseases or syndromes (e.g., bowel obstruction, major GI surgery, short-bowel syndrome, irritable bowel syndrome, inflammatory bowel disease, chronic diarrhea)
* Anemic, defined as a serum hemoglobin concentration <9.0 g/dL
* Inadequate dialysis efficacy, defined as a Kt/V of <1.2
* Dietary restrictions (e.g., allergies) or otherwise unable/unwilling to adhere to study diets (excludes dietary restrictions on high-potassium foods)
* Pregnant or planning to become pregnant during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Pre-dialysis serum potassium concentrations. | Day 1
  Pre-dialysis blood samples will be collected by dialysis center staff, and delivered to the Tisch Laboratory by study staff on each dialysis day.
Pre-dialysis serum phosphorus concentrations. | Day 7
  Post-prandial blood tests will be obtained after the participant consumed the standard meal providing 20% of estimated energy requirements corresponding to the research diet

CONTACTS AND LOCATIONS:
Overall Officials: David St Jules, MD, Principal Investigator — NYU Langone Health